CLINICAL TRIAL: NCT06550297
Title: Enhancing, Culturally Adapting, and Expanding Medically Tailored Meals Programs to Promote Cardiovascular Health Equity
Brief Title: Medically Tailored Meals for Cardiovascular Health
Acronym: MTM4CVH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Nour Makarem, PhD, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAV0681; 24FIM1267661 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Diet, Healthy; HbA1c; Blood Pressure
Keywords: Medically Tailored Meals; Type 2 Diabetes; High Blood Pressure; Multiple Cardiometabolic Morbidity; Food is Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Cohort A (type 2 diabetes patients who currently qualify for MTMs) Active Comparator (Active Comparator): Participants in this arm are type 2 diabetes patients with hypertension or elevated blood pressure who currently qualify for medically tailored meals (MTMs). This arm will receive God's Love We Deliver's current MTM program, which consists of 10 home-delivered MTMs per week and nutritional counseling by a Registered Dietitian Nutritionist for an 8-month period.
  Interventions: Behavioral: Medically Tailored Meals and Nutritional Counseling
- Arm 2: Cohort A (type 2 diabetes patients who currently qualify for MTMs) Intervention (Experimental): Participants in this arm are type 2 diabetes patients with hypertension or elevated blood pressure who currently qualify for medically tailored meals (MTMs). This arm will receive God's Love We Deliver's current MTM program, which consists of 10 home-delivered MTMs per week and nutritional counseling by a Registered Dietitian Nutritionist for an 8-month period (same as Arm 1). In addition, they will receive a culturally and contextually tailored cardiovascular health promotion program that consists of didactic sessions focused on lifestyle change and the American Heart Association's Life's Essential 8 framework, setting weekly specific, measurable, attainable, realistic, and timely (S.M.A.R.T.) goals for health behavior modification, group coaching, cooking demonstrations, recipes and gift bags with healthy ingredients, and addressing social needs.
  Interventions: Behavioral: Medically Tailored Meals and Nutritional Counseling; Behavioral: Cardiovascular Health Promotion Educational Program
- Arm 3: Cohort B (type 2 diabetes patients who do not currently qualify for MTMs) Active Comparator (Active Comparator): Participants in this arm are type 2 diabetes patients with hypertension or elevated blood pressure who do not currently qualify for medically tailored meals (MTM) programs. This arm will receive God's Love We Deliver's current MTM program, which consists of 10 home-delivered MTMs per week and nutritional counseling by a Registered Dietitian Nutritionist for an 8-month period. In addition, they will receive a culturally and contextually tailored cardiovascular health promotion program that consists of didactic sessions focused on lifestyle change and the American Heart Association's Life's Essential 8 framework, setting weekly specific, measurable, attainable, realistic, and timely (S.M.A.R.T.) goals for health behavior modification, group coaching, cooking demonstrations, recipes and gift bags with healthy ingredients, and addressing social needs.
  Interventions: Behavioral: Medically Tailored Meals and Nutritional Counseling; Behavioral: Cardiovascular Health Promotion Educational Program
- Arm 4: Cohort B (type 2 diabetes patients who do not currently qualify for MTMs) Intervention (Experimental): Participants in this arm are type 2 diabetes patients with hypertension or elevated blood pressure who do not currently qualify for medically tailored meals (MTM) programs. This arm will receive the MTM program and nutritional counseling by a Registered Dietitian Nutritionist for an 8-month period but with a distinct MTM dosing schedule. They will receive the regular MTM schedule of 10 MTMs/week for the first 3 months of the intervention. After this initial period, MTM dosing will be gradually reduced by 1 MTM each month to a target schedule of 5 MTMs/week in the final month of the intervention. In addition, they will also receive the same culturally and contextually tailored cardiovascular health promotion program as Arms 2 and 3.
  Interventions: Behavioral: Medically Tailored Meals and Nutritional Counseling; Behavioral: Cardiovascular Health Promotion Educational Program

INTERVENTIONS:
Behavioral: Medically Tailored Meals and Nutritional Counseling — God's Love We Deliver's current MTM program, which consists of weekly home-delivered MTMs and nutritional counseling by a Registered Dietitian Nutritionist for an 8-month period. The Food is Medicine Coalition Clinical Committee establishes and regularly updates the MTM Nutrition Standards, which catalogue the nutrition quality of this evidence-based intervention. Arms 1-3 will receive 10 MTMs per week for 8 months. Arm 4 will receive a distinct dosing down approach as follows: 10 MTMs/week in months 1-3, 9 MTMs/week in month 4, 8 MTMs/week in month 5, 7 MTMs/week in month 6, 6 MTMs/week in month 7, and 5 MTMs/week in month 8.
Behavioral: Cardiovascular Health Promotion Educational Program — Culturally and contextually tailored cardiovascular health promotion program that consists of didactic sessions focused on lifestyle change and the American Heart Association's Life's Essential 8 framework, setting weekly specific, measurable, attainable, realistic, and timely (S.M.A.R.T.) goals for health behavior modification, group coaching, cooking demonstrations, recipes and gift bags with healthy ingredients and fresh produce, and addressing social needs.
  Arms: Arm 2: Cohort A (type 2 diabetes patients who currently qualify for MTMs) Intervention; Arm 3: Cohort B (type 2 diabetes patients who do not currently qualify for MTMs) Active Comparator; Arm 4: Cohort B (type 2 diabetes patients who do not currently qualify for MTMs) Intervention

SUMMARY:
This randomized clinical trial (RCT) will investigate novel approaches to enhance effectiveness, engagement, reach, and cost-effectiveness of medically tailored meals (MTM) programs for promoting cardiovascular health, focusing on economically disadvantaged New York City neighborhoods with a disparate burden of multiple cardiometabolic diseases. The main questions the RCT aims to answer are:

1. Does enhancing MTM programs, with culturally relevant cardiovascular health curriculum (including educational sessions on heart health, healthy diet, cooking demonstrations, recipes, gift bags with healthy ingredients and fresh produce, and addressing social needs) enhance program engagement and effectiveness in improving short-term healthy eating behaviors and clinical outcomes (HbA1c and blood pressure) among individuals with type 2 diabetes and elevated to high blood pressure who currently qualify for MTM programs?
2. Is the MTM program coupled with the cardiovascular health curriculum effective for improving healthy eating behaviors and clinical outcomes (HbA1c and blood pressure) among individuals with type 2 diabetes and elevated to high blood pressure who do not currently qualify for MTM programs and is a gradual reduction of MTM dosing an effective and sustainable approach for expanding reach of these programs?

To answer question 1, 60 participants with type 2 diabetes and elevated to high blood pressure who currently qualify for MTM programs will be randomized into a group that receives the standard MTM program (10 MTMs/week for 8 months) or a group that receives the standard program plus the cardiovascular health curriculum.

To answer question 2, 100 participants with type 2 diabetes and elevated to high blood pressure who do not currently qualify for MTM programs (due to not having advanced disease with complications) will be randomized into a group that receives the standard MTM program (10 MTMs/week for 8 months) plus the cardiovascular health curriculum or a group that receives standard MTM program for the first 3 months followed by a gradual reduction in dosing of the MTMs by 50% over the remaining 5 months plus the CVH curriculum.

All participants will have their HbA1c and blood pressure measured and complete questionnaires about their diet quality, health and lifestyle behaviors, and program engagement and implementation at baseline, 3 months, and 8 months.

DETAILED DESCRIPTION:
Medically tailored meals (MTMs) represent an integral in-kind intervention of the Food Is Medicine (FIM) initiative aimed at providing healthy food in a way that is integrated with the health care sector to prevent and manage chronic disease. MTMs are a promising approach to address diet-related cardiovascular inequities, because they collectively address food and nutrition insecurity, severe illness or chronic cardiometabolic disease, and challenges with activities of daily living such as shopping for or preparing meals in those with complex medical conditions. However, additional research is needed to determine how MTM programs could be enhanced to become more culturally and contextually responsive, increase engagement with these programs, enhance their effectiveness and sustainability, and expand their reach.

ELIGIBILITY:
For Cohort A (Individuals who currently qualify for MTMs)

Inclusion Criteria:

1. Qualifying type 2 diabetes diagnosis (typically physician referred to the program due to more advanced disease with uncontrolled diabetes and complications)
2. Hypertension diagnosis (systolic blood pressure greater than or equal to 130 mmHg and/or diastolic blood pressure greater than or equal to 80 mmHg) or elevated blood pressure (defined as systolic blood pressure greater than or equal to 120 mmHg)

Exclusion Criteria:

1. Cancer diagnosis
2. Undergoing cancer treatment
3. Non-English or non-Spanish speaking
4. Not cognitively able to complete study requirements
5. Severe psychiatric disorders
6. Inability to provide informed consent
7. Health conditions that could prevent safe participation or impact study outcomes (e.g., substance use disorder, dialysis, neurodegenerative conditions)

For Cohort B (Individuals who do not currently qualify for MTMs)

Inclusion Criteria:

1. Type 2 diabetes diagnosis (physician diagnosed or HbA1c greater than or equal to 6.5% or diabetes medication use)
2. Hypertension diagnosis (systolic blood pressure greater than or equal to 130 mmHg and/or diastolic blood pressure greater than or equal to 80 mmHg or physician diagnosis or hypertension medication use) or elevated blood pressure (defined as systolic blood pressure greater than or equal to 120 mmHg)

Exclusion Criteria:

1. Cancer diagnosis
2. Undergoing cancer treatment
3. Non-English or non-Spanish speaking
4. Not cognitively able to complete study requirements
5. Severe psychiatric disorders
6. Inability to provide informed consent
7. Health conditions that could prevent safe participation or impact study outcomes (e.g., substance use disorder, dialysis, neurodegenerative conditions)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Diet Quality | baseline to 8 months
  The Mediterranean Eating Pattern for Americans (MEPA) scale, which captures adherence to a heart healthy dietary pattern, will be used to assess diet quality. The MEPA score ranges from 0-16 with higher scores indicating better diet quality. The change in MEPA scores from baseline to 8 months will be calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Mean Diet Quality | baseline to 8 months
  The Mediterranean Eating Pattern for Americans (MEPA) scale, which captures adherence to a heart healthy dietary pattern, will be used to assess diet quality. The MEPA score ranges from 0-16 with higher scores indicating better diet quality. The mean MEPA scores at 8 months will be calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).

SECONDARY OUTCOMES:
Change in Diet Quality (Interim Change at 3 months) | baseline, 3 months
  The Mediterranean Eating Pattern for Americans (MEPA) scale, which captures adherence to a heart healthy dietary pattern, will be used to assess diet quality. The MEPA score ranges from 0-16 with higher scores indicating better diet quality. The change in MEPA scores from baseline to 3 months will be calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Mean Diet Quality (Interim at 3 months) | baseline, 3 months
  The Mediterranean Eating Pattern for Americans (MEPA) scale, which captures adherence to a heart healthy dietary pattern, will be used to assess diet quality. The MEPA score ranges from 0-16 with higher scores indicating better diet quality. The mean MEPA scores at 3 months will be calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Change in HbA1c | baseline, 3 months, 8 months
  A fast and accurate HbA1c fingerstick test will assess changes in glycemic control from baseline to 3 months and 8 months (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Mean HbA1c | baseline, 3 months, 8 months
  A fast and accurate HbA1c fingerstick test will assess glycemic control and mean HbA1c will be compared at 3 months and 8 months (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Change in systolic blood pressure | baseline, 3 months, 8 months
  The change office systolic blood pressure (mmHg) from baseline to follow-up at 3 months and 8 months will be calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Change in diastolic blood pressure | baseline, 3 months, 8 months
  The change office diastolic blood pressure (mmHg) from baseline to follow-up at 3 months and 8 months will be calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Mean systolic blood pressure | baseline, 3 months, 8 months
  Mean office systolic blood pressure (mmHg) at 3 months (mid-trial) and 8-months of follow-up (end of trial) calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Mean diastolic blood pressure | baseline, 3 months, 8 months
  Mean office diastolic blood pressure (mmHg) at 3 months (mid-trial) and 8-months of follow-up (end of trial) calculated and compared across randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Acceptability of Implementation | 8 months
  Acceptability will be measured by questionnaire. Items are adapted from the validated Acceptability of Implementation Measure (AIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better intervention acceptability. The items are analyzed individually and not summed to a total score.
Feasibility of Implementation | 8 months
  Feasibility will be measured by questionnaire using items adapted from the validated Feasibility of Implementation Measure (FIM) and rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better feasibility. The items are analyzed individually and not summed to a total score.
Appropriateness of Implementation | 8 months
  Appropriateness will be measured by questionnaire. Items are adapted from the validated Implementation Appropriateness Measure (IAM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better appropriateness. The items are analyzed individually and not summed to a total score.
Satisfaction with Intervention | 8 months
  Satisfaction with the intervention components will be measured by questionnaire. Participants will rate their satisfaction with intervention by indicating how likely they are to recommend it to others on a 10-point scale with higher scores indicating greater satisfaction. They will also be asked to rate the quality of the intervention as poor, fair, good, very good, or excellent. The items are analyzed individually and not summed to a total score.

OTHER OUTCOMES:
Food Insecurity | baseline, 3 month, 8 months
  The USDA Household Food Security Survey (FSSM-6 item) will be administered at baseline, 3 months, and 8 months. The scores range from 0-6 such that a score of 0-1 indicates high or marginal food security, 2-4 indicates low food security, and 5-6 indicates very low food security. Changes in the score from baseline to follow up at 3 month and 8 months will be evaluated. In addition differences in mean scores will be compared across the randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Nutrition Insecurity | baseline, 3 months, 8 months
  The Gretchen Swanson 4-item nutrition screener will be administered at baseline, 3 months, and 8 months (score range: 0-4 with higher scores indicating higher nutrition security). Changes in the score from baseline to follow up at 3 month and 8 months will be evaluated. In addition differences in mean scores will be compared across the randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Sleep Health | baseline, 3 month, 8 months
  Sleep duration and quality will be measured using the Pittsburgh Sleep Quality Index (PSQI, score range: 0-21). Changes in self-reported habitual hours of sleep and the PSQI score from baseline to follow up at 3 month and 8 months will be evaluated. In addition differences in mean sleep duration and PSQI scores will be compared across the randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
Self-rated health | baseline, 3 months, 8 months
  Participant will rate their health as excellent, very good, good, fair, or poor at baseline, 3 months, and 8 months. Changes in self-rated health from baseline to follow up at 3 month and 8 months as well as the differences in mean self-rated health will be compared across the randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).
General Health Status | baseline, 3 month, 8 months
  The EuroQoL 5-Dimension 5-Level (EQ-5D-5L) will be used to measure general health status and quality of life. This will be captured based on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Based on the participant's response for reach dimension they will receive a 1-digit number, and the digits for the five dimensions will be combined into a 5-digit number that describes the patient's health state. This study will evaluate changes in this measure from baseline to follow up at 3 month and 8 months. In addition, differences in mean scores will be compared across the randomization arms (comparing Arm 1 vs. Arm 2 and Arm 3 vs. Arm 4).

CONTACTS AND LOCATIONS:
Overall Officials: Nour Makarem, PhD, FAHA, Principal Investigator — Columbia University
Locations (1):
- Columbia University Mailman School of Public Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared de-identified and in aggregate, consistent with the American Hospital Association Healthcare x Food requirements.